CLINICAL TRIAL: NCT00005007
Title: Wegener's Granulomatosis Etanercept Trial (WGET)
Brief Title: Etanercept for Wegener's Granulomatosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: John H. Stone, M.D., M.P.H., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01 AR92240; NIAMS-041
Record Dates: First submitted 2000-03-24; First posted 2000-03-27 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Wegener's Granulomatosis
Keywords: Wegener's granulomatosis; Vasculitis; Etanercept; Tumor necrosis factor
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Vasculitis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
This study will determine if the drug etanercept, also called Enbrel, is effective in producing and maintaining remission (reduction of disease symptoms) of Wegener's granulomatosis (WG). Etanercept blocks the action of tumor necrosis factor-alpha, a substance that may be involved in inflammatory conditions such as WG. Eight clinical centers around the United States will enroll 181 people who have WG. Patients will have an equal chance to receive either etanercept or placebo (inactive treatment). We will treat patients with standard medications for WG in addition to either etanercept or placebo. We will treat all patients with tapering doses of corticosteroids.

After the patients' disease is controlled (in remission), we will reduce the dosages of the standard medications to lower the risk of side effects associated with these drugs. During the study, we will collect and save blood and tissues samples from patients and use the samples to address other medical questions, such as the cause of WG and factors that lead to disease progression.

DETAILED DESCRIPTION:
The Wegener's Granulomatosis Etanercept Trial (WGET) is a randomized, placebo-controlled clinical trial. A primary objective of the trial is to evaluate the safety and efficacy of etanercept (Enbrel; Immunex Corporation, Seattle, WA) for the induction and maintenance of disease remissions for people with Wegener's granulomatosis (WG) when used in conjunction with standard medications. A secondary objective is to develop a specimen bank of serum, plasma, whole blood, and tissue biopsy samples that may be used to address basic questions regarding the etiology, pathophysiology, and monitoring of WG.

The trial is a phase II/III randomized, double-masked, multicenter trial with a parallel treatment design. We will assign patients randomly to either etanercept or placebo in an assignment ratio of 1:1. In addition to either etanercept or placebo, we will treat all patients with standard drug regimens for WG according to the severity of their disease. We will treat those with limited WG with methotrexate and corticosteroids, and those with severe WG with cyclophosphamide and corticosteroids. After the patients' disease is controlled with therapy (i.e., the standard treatment regimen plus either etanercept or placebo), we will taper the standard medications according to regimens designed to ensure patient safety, diminish morbidity associated with the standard medications, and test the efficacy of etanercept in sustaining disease remissions.

The principal outcome measure in this trial is the number of patients in the two treatment arms who achieve sustained remissions measured by the Birmingham Vasculitis Activity Score for WG (BVAS). The sample size is 181 patients recruited at eight clinical centers in the United States. We will stratify randomization by clinic and disease severity (limited versus severe). Every patient enrolled will have a BVAS of at least three, insuring unequivocally active disease.

We will follow all randomized patients, regardless of whether or not they remain on their assigned treatments, until the common closing date of the trial, defined as 12 months after enrollment of the last patient. We will perform the primary analyses on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum weight of 40 kg.
* Diagnosis of WG, excluding infections, malignancies, systemic autoimmune disorders, and other forms of vasculitis that may mimic WG.
* At least two of the five modified American College of Rheumatology (ACR) criteria for a diagnosis of WG. The modified ACR criteria are: (1) nasal or oral inflammation, defined as the development of painful or painless oral ulcers or purulent or bloody nasal discharge; (2) abnormal chest radiograph, defined as the presence of nodules, fixed infiltrates, or cavities; (3) active urinary sediment, defined as microscopic hematuria (> 5 red blood cells per high-power field) or red blood cell casts; (4) granulomatous inflammation on biopsy, defined as histologic changes showing granulomatous inflammation within the wall of an artery or in the perivascular or extravascular area (artery or arteriole); and (5) positive serum ELISA for ANCAs (anti-neutrophil cytoplasmic antibodies) directed at PR-3.
* Birmingham Vasculitis Activity Score (BVAS) score 3 or greater within 28 days of randomization. This may include either the presence of one or more major items (3 points each) or the presence of three or more minor items (1 point each).
* Willingness and ability, with the assistance of a caregiver if necessary, to comply with treatment and followup procedures.
* Willingness of men and women of childbearing potential to practice an adequate method of birth control during the study and for 3 months afterwards.
* Willingness to limit alcohol consumption to one alcoholic drink per week while taking methotrexate.
* Willingness to refrain from breast-feeding during the study and for 3 months afterwards.
* Collection of all baseline data within 14 days prior to randomization.
* Signed consent statement.

Exclusion Criteria:

* Presence of an active systemic infection.
* White blood cell count less than 4,000/mm cubed or a platelet count less than 120,000/mm cubed.
* Creatinine greater than 2.0 mg/dL secondary to non-WG causes (e.g., hypertensive nephropathy) for a patient with limited disease.
* Known acute or chronic liver disease.
* History of multiple sclerosis or other neurological symptoms suggesting a demyelinating syndrome.
* Current evidence of malignancy or malignancy diagnosed within 5 years of study entry. Patients with squamous or basal cell carcinomas of the skin may be enrolled if they have received curative surgical treatment.
* Positive serum pregnancy test for women of childbearing potential.
* Previous treatment with specific therapies directed against tumor necrosis factor, e.g., etanercept or infliximab.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181
Dates: Start 2000-06; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Number of patients in the two treatment arms who achieve sustained remissions as measured by the Birmingham Vasculitis Activity Score (BVAS) for WG | Measured at study completion

CONTACTS AND LOCATIONS:
Overall Officials: John H. Stone, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Beth Israel Medical Center, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Stone JH, Uhlfelder ML, Hellmann DB, Crook S, Bedocs NM, Hoffman GS. Etanercept combined with conventional treatment in Wegener's granulomatosis: a six-month open-label trial to evaluate safety. Arthritis Rheum. 2001 May;44(5):1149-54. doi: 10.1002/1529-0131(200105)44:53.0.CO;2-F. PMID 11352248
- [Background] Stone JH, Hoffman GS, Merkel PA, Min YI, Uhlfelder ML, Hellmann DB, Specks U, Allen NB, Davis JC, Spiera RF, Calabrese LH, Wigley FM, Maiden N, Valente RM, Niles JL, Fye KH, McCune JW, St Clair EW, Luqmani RA; International Network for the Study of the Systemic Vasculitides (INSSYS). A disease-specific activity index for Wegener's granulomatosis: modification of the Birmingham Vasculitis Activity Score. International Network for the Study of the Systemic Vasculitides (INSSYS). Arthritis Rheum. 2001 Apr;44(4):912-20. doi: 10.1002/1529-0131(200104)44:43.0.CO;2-5. PMID 11318006
- [Background] WGET Research Group. Design of the Wegener's Granulomatosis Etanercept Trial (WGET). Control Clin Trials. 2002 Aug;23(4):450-68. doi: 10.1016/s0197-2456(02)00209-x. PMID 12161090
- [Result] Stone JH; Wegener's Granulomatosis Etanercept Trial Research Group. Limited versus severe Wegener's granulomatosis: baseline data on patients in the Wegener's granulomatosis etanercept trial. Arthritis Rheum. 2003 Aug;48(8):2299-309. doi: 10.1002/art.11075. PMID 12905485
- [Result] Merkel PA, Lo GH, Holbrook JT, Tibbs AK, Allen NB, Davis JC Jr, Hoffman GS, McCune WJ, St Clair EW, Specks U, Spiera R, Petri M, Stone JH; Wegener's Granulomatosis Etanercept Trial Research Group. Brief communication: high incidence of venous thrombotic events among patients with Wegener granulomatosis: the Wegener's Clinical Occurrence of Thrombosis (WeCLOT) Study. Ann Intern Med. 2005 Apr 19;142(8):620-6. doi: 10.7326/0003-4819-142-8-200505030-00011. PMID 15838068
- [Result] Stone JH, Rajapakse VN, Hoffman GS, Specks U, Merkel PA, Spiera RF, Davis JC, St Clair EW, McCune J, Ross S, Hitt BA, Veenstra TD, Conrads TP, Liotta LA, Petricoin EF 3rd; Wegener's Granulomatosis Etanercept Trial Research Group. A serum proteomic approach to gauging the state of remission in Wegener's granulomatosis. Arthritis Rheum. 2005 Mar;52(3):902-10. doi: 10.1002/art.20938. PMID 15751091
- [Result] Seo P, Min YI, Holbrook JT, Hoffman GS, Merkel PA, Spiera R, Davis JC, Ytterberg SR, St Clair EW, McCune WJ, Specks U, Allen NB, Luqmani RA, Stone JH; WGET Research Group. Damage caused by Wegener's granulomatosis and its treatment: prospective data from the Wegener's Granulomatosis Etanercept Trial (WGET). Arthritis Rheum. 2005 Jul;52(7):2168-78. doi: 10.1002/art.21117. PMID 15986348
- [Result] Wung PK, Holbrook JT, Hoffman GS, Tibbs AK, Specks U, Min YI, Merkel PA, Spiera R, Davis JC, St Clair EW, McCune J, Ytterberg SR, Allen NB, Stone JH; WGET Research Group. Herpes zoster in immunocompromised patients: incidence, timing, and risk factors. Am J Med. 2005 Dec;118(12):1416. doi: 10.1016/j.amjmed.2005.06.012. PMID 16378799
- [Result] Stone JH, Holbrook JT, Marriott MA, Tibbs AK, Sejismundo LP, Min YI, Specks U, Merkel PA, Spiera R, Davis JC, St Clair EW, McCune WJ, Ytterberg SR, Allen NB, Hoffman GS; Wegener's Granulomatosis Etanercept Trial Research Group. Solid malignancies among patients in the Wegener's Granulomatosis Etanercept Trial. Arthritis Rheum. 2006 May;54(5):1608-18. doi: 10.1002/art.21869. PMID 16646004
- [Derived] Clowse ME, Copland SC, Hsieh TC, Chow SC, Hoffman GS, Merkel PA, Spiera RF, Davis JC Jr, McCune WJ, Ytterberg SR, St Clair EW, Allen NB, Specks U, Stone JH; WGET Research Group. Ovarian reserve diminished by oral cyclophosphamide therapy for granulomatosis with polyangiitis (Wegener's). Arthritis Care Res (Hoboken). 2011 Dec;63(12):1777-81. doi: 10.1002/acr.20605. PMID 22127969